CLINICAL TRIAL: NCT01401049
Title: Preventing Propofol Injection Pain: Prospective Randomized Trial Comparing Propofol Versus Fospropofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-0742
Record Dates: First submitted 2011-06-17; First posted 2011-07-25 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Complication of Injection; Pain
Keywords: Fospropofol; Propofol; Colonoscopy; Lusedra
MeSH Terms: conditions — Pain | interventions — fospropofol; Propofol; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fospropofol (Experimental): To compare the incidence and intensity of pain on injection that is caused by propofol (lipid emulsion) versus the test drug fospropofol. A third arm will also be included using a current standard (propofol plus lidocaine) as a methodological control.
  Interventions: Drug: Fospropofol
- Propofol/Lidocaine (Active Comparator): The purpose of this study is to compare the incidence and intensity of possible pain on injection as well as patient satisfaction caused by propofol (a lipid based medication); Lusedra (a water based medication); and the drug combination of propofol with lidocaine (a local anesthetic commonly used with propofol injection).
  Interventions: Drug: Propofol/Lidocaine

INTERVENTIONS:
Drug: Fospropofol — To compare the incidence and intensity of pain on injection that is caused by propofol (lipid emulsion) versus the test drug fospropofol. A third arm will also be included using a current standard (propofol plus lidocaine) as a methodological control.
  Arms: Fospropofol
Drug: Propofol/Lidocaine — We plan to assess the incidence and intensity of pain on injection that is caused by propofol (lipid emulsion).
  Other Names: Propofol; Fospropofol; Pain on Injection
  Arms: Propofol/Lidocaine

SUMMARY:
The purpose of this study is to compare the incidence and intensity of possible pain on injection as well as patient satisfaction caused by propofol (a lipid based medication); Lusedra (a water based medication); and the drug combination of propofol with lidocaine (a local anesthetic commonly used with propofol injection).

DETAILED DESCRIPTION:
Propofol (2,6-diisopropylphenol) is one of the most common induction and sedative agents used today. Properties that make this agent popular include rapid onset and quick recovery. However, as its use became more widespread, side effects such as pain on injection have attracted more attention. The incidence of pain on propofol injection is as high as 70 - 90%. Numerous studies report that more than 50% of patients recall the unpleasant burning sensation during injection.

Many techniques to minimize pain on injection associated with propofol have been described; pre-administration of different medications including lidocaine, ketamine, thiopental, metoclopramide, dexamethasone, ondansetron, and remifentanil have been reported with mixed success. Some have even tried to use lidocaine with a tourniquet. Others have reported the use of distraction techniques including counting numbers aloud.

Recently, a solvent mixture of medium chain triglyceride and long chain triglyceride has been tested for prevention of pain on propofol injection. Lusedra (fospropofol disodium), the water-soluble prodrug of propofol, does not cause pain on injection as it is water based medication. Demonstrating the benefit of fospropofol over propofol in patient satisfaction will improve acceptance by anesthesia providers.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I, II or III.
* Age 18 - 65.
* Both male and female.
* No significant laboratory abnormalities.

Exclusion Criteria:

* Chronic pain patients or patients receiving benzodiazepines or opioids / other analgesics for control of acute pain will be excluded.
* Patients with known allergies to any of the study drugs, or to soybean oil or egg lecithin are excluded.
* Women with a positive pregnancy test reported from pre-surgical testing or their physician's office or who are breast feeding at the time of surgery.
* No emergency patients will be recruited for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Lee, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Tisch Hospital, part of New York University (NYU) Langone Medical Center. An additional site was opened, Research Associates of New York (RANY). All patients having either a colonoscopy or upper endoscopy, or both, were considered.
Period: Overall Study
Arm/Group | Fospropofol | Propofol/Lidocaine
Started | 0 (Due to flooding from Hurricane Sandy at our site, all files and pertinent patient data were lost.) | 0 (Due to flooding from Hurricane Sandy at our site, all files and pertinent patient data were lost.)
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to flooding from Hurricane Sandy at our site, all files and pertinent patient data were lost.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fospropofol | Propofol/Lidocaine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Compare Incidence and Intensity of Pain on Injection That is Caused by Propofol (Lipid Emulsion) Versus the Test Drug Fospropofol.
Description: We hypothesize that we can reject the null hypothesis that results from all 3 arms are from the same sample, and then show (in pair wise tests) that fospropofol is superior to propofol, and not-inferior to propofol plus lidocaine.
Time Frame: 2 hours
Population: Due to flooding from Hurricane Sandy at our site, all files and pertinent patient data were lost.
Arm/Group | Fospropofol | Propofol/Lidocaine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Compare Patient Satisfaction With Sedation Including the Recall of Pain.
Description: as for outcome 1
Time Frame: 2 hours after the end of the procedure.
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Fospropofol | Propofol/Lidocaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fospropofol | Propofol/Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No